CLINICAL TRIAL: NCT04054154
Title: Pilot Study to Evaluate the Feasibility of Measuring (a) Intratumoral Pressures Using a Novel Piezo- Resistive Semiconductor Catheter and (b) Intratumoral Stiffness Using Shear Wave Elastography With Ultrasound
Brief Title: An Investigational Device (Millar Mikro-Tip Catheter) and Imaging Scan (Shear Wave Elastography) in Measuring Tumor Pressure and Stiffness in Patients With Solid Tumors Undergoing Ultrasound-Guided Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014-0038; NCI-2019-02647 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0038 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-28; First posted 2019-08-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-01

CONDITIONS: Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device Feasibility (Millar Mikro-tip catheter, elastography) (Experimental): Patients scheduled for an ultrasound-guided tumor biopsy undergo stiffness assessment of the tumor with shear wave elastography over 2 minutes and pressure measurements of the tumor using a Millar Mikro-tip catheter before and after the biopsy is collected.
  Interventions: Device: Shear Wave Elastography; Procedure: Tumor Interstitial Fluid Pressure Measurement

INTERVENTIONS:
Device: Shear Wave Elastography — Undergo shear wave elastography
  Other Names: Transient Elastography
Procedure: Tumor Interstitial Fluid Pressure Measurement — Undergo tumor pressure measurement

SUMMARY:
This trial studies how well a Millar Mikro-tip catheter and shear wave elastography measure pressure and stiffness inside tumors among patients with solid tumors undergoing an ultrasound-guided biopsy. A Millar Mikro-tip catheter measures the pressure inside the tumor. Shear wave elastography is similar to an ultrasound and uses sound waves to vibrate the tissue in order to study tissue stiffness. These measurements may help doctors learn if pressure and stiffness are related to intratumoral fibrosis (the thickening and scarring of connective tissue).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of measuring tumor intratumoral pressures in vivo using a commercially available, sterile, single use, cardiovascular catheter device.

II. To determine the feasibility of measuring tumor intratumoral stiffness in vivo using a commercially available shear wave elastography with ultrasound.

SECONDARY OBJECTIVES:

I. To assess the relationship of tumor pressure, stiffness, and fibrosis.

OUTLINE:

Patients scheduled for an ultrasound-guided tumor biopsy undergo stiffness assessment of the tumor with shear wave elastography over 2 minutes and pressure measurements of the tumor using a Millar Mikro-tip catheter before and after the biopsy is collected.

After completion of the study, patients are followed up at 24-48 hours and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for at least one biopsy (diagnostic or research) for solid organ tumors (excluding bone) at MD Anderson.
* Patients who are able to understand and give consent to participation in the study.

Exclusion Criteria:

* Tumor size < 1.5 cm or > 5 cm in size on pre-procedural imaging for 1st assessment and < 1 cm for 2nd assessment
* Pregnant women (these patients will be tested for pregnancy before they are scheduled for a diagnostic or research biopsy per inclusion criteria #1).
* Tumors involving bone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
The change in Tumor pressure | Up to 30 days
  Measured by Millar Microcath (Millar Mikro-Tip Pressure Catheter). Tumor pressure and its change will be summarized using mean, standard deviation, and range by time point.
The change in Tumor stiffness | Up to 30 days
  Measured by General Electric LOGIQ Shear Wave Elastography. Tumor stiffness and its change will be summarized using mean, standard deviation, and range by time point.

SECONDARY OUTCOMES:
Tumor pressure | Up to 30 days
  As a secondary endpoint, the relationship of tumor pressure with tumor fibrosis will be assessed for each patient. An ordinary least squares regression will be fit to the data to investigate the potential relationship between tumor stiffness, pressure, and fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Y Huang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT04054154/ICF_000.pdf